CLINICAL TRIAL: NCT02228031
Title: The Influence of Oxytocin on the Mirror Neuron System: Developing Brain Imaging Paradigms for Future Therapeutic Interventions
Brief Title: Oxytocin, Emotions and Mirror Neurons
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: University of Maryland, College Park (Other)
Responsible Party: Principal Investigator, Robert Buchanan, Interim Director, Maryland Psychiatric Research Center, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: HP-00059904
Record Dates: First submitted 2014-08-15; First posted 2014-08-28 (Estimated); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Social Cognition; Expressed Emotion
Keywords: Mirror neurons; Imitation; Oxytocin
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Oxytocin (Experimental): The experimental oxytocin group will receive 24 international units (IU) of oxytocin using an intranasal administration (self-administered nasal spray) one time before the experimental session.
  Interventions: Drug: Oxytocin
- Placebo (Placebo Comparator): The placebo comparator group will receive sterile saline through intranasal administration, consisting of the same salt solution in which the hormone will be dissolved , but lacking the hormone itself.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Oxytocin — The experimental oxytocin group will receive 24 international units (IU) of oxytocin using an intranasal administration (self-administered nasal spray) one time before the experimental session
  Other Names: Syntocinon nasal spray
  Arms: Oxytocin
Other: Placebo — The placebo comparator group will receive sterile saline through intranasal administration, consisting of the same salt solution in which the hormone will be dissolved , but lacking the hormone itself.
  Arms: Placebo

SUMMARY:
The purpose of this project is to investigate the possible effect of intranasally administered Oxytocin (OT) on specific mirror neuron areas in human brain. The mirror neuron system (MNS) is thought to be involved in action perception and understanding, and may also underlie more complex cognitive processes such as imitation. We will use electroencephalographic (EEG) investigations to examine brain activity while participants complete two different tasks, consisting of the observation and imitation of emotional facial expressions (video presented) and the observation and execution of simple grasping actions (live presented), respectively. In addition, before the beginning of the EEG recording session, subjects will be randomly assigned to two different groups (Oxytocin or Placebo group) and will receive a dose of either intranasal Oxytocin or Placebo solution. Oxytocin is a polypeptide hormone that plays a critical role in social behavior. We will identify mu and beta rhythm from the ongoing EEG and examine suppression as a function of emotion and goal directed action perception and imitation/execution.

ELIGIBILITY:
Inclusion Criteria:

* Right-hand dominant
* Sufficient spoken English so as to be able to complete testing validly and give informed consent

Exclusion Criteria:

* Currently taking any psychotropic or cognition enhancing medication
* History of schizophrenia or any other psychotic disorder, including Bipolar Disorder
* Family history of psychosis
* Neurological disease or clinically significant head injury
* Physical disability that substantially impairs motor function
* Current diagnosis of polydypsic-induced hyponatremia
* Substance dependence or abuse in the past 6 months

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
EEG mu rhythm suppression | Before oxytocin/placebo administration and 45 minutes after
  The EEG mu rhythm suppression is an index of the human mirror neuron system (alpha and lower beta band activity (8-13 and ~20Hz) recorded over the sensorimotor cortex. EEG will be recorded during the performance of an emotion imitation task (Carr et al., 2003) in which participants will be asked to imitate and internally generate facial emotions seen on a computer screen, or to simply observe, as well as performing a simple grasping action task. Changes in the mu suppression while the performance of these tasks, before and after oxytocin/placebo administration, will be the primary outcome measure.

CONTACTS AND LOCATIONS:
Overall Officials: Robert W Buchanan, MD, Principal Investigator — University of Maryland, College Park; Nathan Fox, PhD, Study Director — University of Maryland, College Park
Locations (1):
- Child Development Lab, University of Maryland, College Park, Maryland, United States

REFERENCES:
- [Background] Carr L, Iacoboni M, Dubeau MC, Mazziotta JC, Lenzi GL. Neural mechanisms of empathy in humans: a relay from neural systems for imitation to limbic areas. Proc Natl Acad Sci U S A. 2003 Apr 29;100(9):5497-502. doi: 10.1073/pnas.0935845100. Epub 2003 Apr 7. PMID 12682281